CLINICAL TRIAL: NCT05038969
Title: Comparative Randomized, Single Dose,Two-way Crossover Bioequivalence Study to Determine the Bioequivalence of Esomeprazole From Stomopral 40 mg Capsules Contain Enteric Coated Pellets (Future Pharmaceuticals Industries, Egypt) and Nexium 40 mg Delayed Release Capsules (AstraZeneca Sweden, Product of France)
Brief Title: Bioequivalence Study of Esomeprazole From Stomopral 40 mg Capsules Contain Enteric Coated Pellets (Future Pharmaceuticals Industries, Egypt) and Nexium 40 mg Delayed Release Capsules (AstraZeneca Sweden, Product of France)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genuine Research Center, Egypt (Industry)
Collaborators: Future Pharmaceuticals Industries, Egypt (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GRC/1/20/868
Record Dates: First submitted 2021-09-06; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Healthy
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A test (Experimental): Test drug (Stomopral) 1 capsule contains 40 mg Enteric Coated Pellets of Esomeprazole
  Interventions: Drug: Stomopral
- B reference (Active Comparator): Reference drug (Nexium) 1 capsule contains 40 mg Esomeprazole
  Interventions: Drug: Nexium

INTERVENTIONS:
Drug: Stomopral — 1 capsule contains 40 mg Esomeprazole
  Other Names: Nexium
  Arms: A test
Drug: Nexium — 1 capsule contains 40 mg Esomeprazole
  Arms: B reference

SUMMARY:
Comparative randomized, single dose Bioequivalence Study of Esomeprazole From Stomopral 40 mg Capsules Contain Enteric Coated Pellets (Future Pharmaceuticals Industries, Egypt) and Nexium 40 mg Delayed Release Capsules (AstraZeneca Sweden, Product of France) in Healthy Human Volunteers Under Fasting Condition.

DETAILED DESCRIPTION:
Healthy volunteers, 18-55 years of age, selected from the Egyptian population fulfilling the selection criteria. Minimum of 24 subjects will participate in the study. All dosed subject samples will be analyzed and their data will be included in the final study report.

Primary Pharmacokinetic Parameters: Cmax, AUC0→t and AUC0→∞ Secondary Pharmacokinetic Parameters: Ke, tmax and t1/2e. ANOVA using 5% significance level for transformed (with the 90% confidence intervals) and untransformed data of Cmax, AUC0-72 and AUC0-∞ for untransformed data of Ke, tmax and t1/2e.

The confidence intervals of logarithmically transformed Test/Reference ratios for Cmax, AUC0-72 and AUC0-∞ to be within 80.00-125.00%.

A comprehensive final report will be issued upon the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, age 18 to 55 years, inclusive.
2. Body weight within 15% of normal range according to the accepted normal values for body mass index (BMI).
3. Medical demographics without evidence of clinically significant deviation from normal medical condition, eg.: no history of heart, liver, kidney, gastrointestinal, nervous system, or metabolic abnormalities.
4. Results of clinical laboratory test are within the normal range or with a deviation that is not considered clinically significant by principal investigator.
5. Females should be on a suitable birth control method.
6. Fully informed subjects that consented to participate in the study.

Exclusion Criteria:

1. Subjects with known allergy to the products tested.
2. Female subjects who were pregnant or nursing.
3. Acute infection within one week preceding first study drug administration.
4. History of drug or alcohol abuse.
5. Subject does not comply with the stated instruction of not taking any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.
6. Subject is on a special diet (for example subject is vegetarian).
7. Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.
8. Subject does not agree not to consume any beverages or foods containing grapefruit 7 days prior to first study drug administration until the end of the study.
9. Subject has a family history of severe diseases which have direct impact on the study.
10. Participation in a bioequivalence study or in a clinical study within the last 8 weeks before first study drug administration.
11. Subject intends to be hospitalized within 3 months after first study drug administration.
12. Subjects who has blood donated or lost more than 500 mL blood within 3 months prior to the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Cmax | Up to12 hours post dose in each treatment period
  Maximal measured plasma concentration

SECONDARY OUTCOMES:
Time of the maximum plasma concentration (Tmax) | Up to12 hours post dose in each treatment period
  The amount of time that a drug is present at the maximum concentration in serum

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshafeey, Ph.D. Pharma, Study Director — Genuine Research Center
Locations (1):
- Genuine Research Center GRC, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow SC, Wang H. On sample size calculation in bioequivalence trials. J Pharmacokinet Pharmacodyn. 2001 Apr;28(2):155-69. doi: 10.1023/a:1011503032353. PMID 11381568
- [Background] Diletti E, Hauschke D, Steinijans VW. Sample size determination for bioequivalence assessment by means of confidence intervals. Int J Clin Pharmacol Ther Toxicol. 1991 Jan;29(1):1-8. PMID 2004861
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848